CLINICAL TRIAL: NCT01516957
Title: A Randomized, Double-blinded, Placebo-controlled, Multiple-dose Study With an Open Label Extension to Evaluate the Safety and Efficacy of AMG 827 in Subjects With Psoriatic Arthritis.
Brief Title: AMG 827 in Subjects With Psoriatic Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20101227
Record Dates: First submitted 2011-08-18; First posted 2012-01-25 (Estimated); Results first posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; IL-17; AMG 827; AMG827; Musculoskeletal Disease; Spondylarthropathy
MeSH Terms: conditions — Arthritis, Psoriatic; Musculoskeletal Diseases; Spondylarthropathies

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- AMG 827 140 (Experimental): 140 mg AMG 827
  Interventions: Drug: AMG 827 140
- Placebo SC (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- AMG 827 280 (Experimental): 280 mg AMG 827
  Interventions: Drug: AMG 827 280
- AMG 827 210 (Experimental): AMG 827 SC 210 mg
  Interventions: Drug: AMG 827 210

INTERVENTIONS:
Drug: AMG 827 140 — 140 mg AMG 827 SC (subcutaneous)
  Arms: AMG 827 140
Drug: Placebo — Placebo SC (subcutaneous)
  Arms: Placebo SC
Drug: AMG 827 280 — 280 mg AMG 827 SC (subcutaneous)
  Arms: AMG 827 280
Drug: AMG 827 210 — 210 mg AMG 827 SC (subcutaneous)
  Arms: AMG 827 210

SUMMARY:
The study will examine the safety and effectiveness of AMG 827 for the treatment of psoriatic arthritis

DETAILED DESCRIPTION:
The study will examine the safety and effectiveness of AMG 827 for the treatment of psoriatic arthritis. Patients will randomly receive either AMG 827 or placebo (a look-a-like liquid that does not have any drug in it) and neither the doctor nor the patient will know what treatment is being given.

ELIGIBILITY:
Inclusion Criteria:

* Subject has had a diagnosis of psoriatic arthritis (by the Classification of Psoriatic Arthritis (CASPAR) criteria) for at least 6 months
* Subject has ≥ 3 tender and ≥ 3 swollen joints

Exclusion Criteria:

* Subject has an active infection or history of infections (systemic anti-infectives were used within 28 days; requiring hospitalization or intravenous anti-infectives within 8 weeks; recurrent or chronic)
* Significant concurrent medical conditions
* Pregnant or breast feeding
* Significant Laboratory abnormalities
* Use of sulfasalazine, hydroxychloroquine, systemically administered calcineurin inhibitors, azathioprine, parenteral corticosteroids including intramuscular or intraarticular administration, or live vaccines within 28 days
* Use of anti-TNF therapy within 2 months
* Use of an anti-interleukin (IL)12/IL-23 drug or other experimental or commercially available biologic therapies for psoriasis and/or psoriatic arthritis within 3 months
* Prior use of rituximab
* Prior use of anti-IL-17 biologic therapy, including AMG 827

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (30):
- United States (22):
  - Research Site, Peoria, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Hemet, California
  - Research Site, Huntington Beach, California
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Palm Desert, California
  - Research Site, Palo Alto, California
  - Research Site, Victorville, California
  - Research Site, Sarasota, Florida
  - Research Site, Boise, Idaho
  - Research Site, Lexington, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Frederick, Maryland
  - Research Site, Grand Rapids, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Lebanon, New Hampshire
  - Research Site, Rochester, New York
  - Research Site, Portland, Oregon
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Seattle, Washington
- Canada (8):
  - Research Site, Victoria, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Newmarket, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Québec

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Mease PJ, Genovese MC, Greenwald MW, Ritchlin CT, Beaulieu AD, Deodhar A, Newmark R, Feng J, Erondu N, Nirula A. Brodalumab, an anti-IL17RA monoclonal antibody, in psoriatic arthritis. N Engl J Med. 2014 Jun 12;370(24):2295-306. doi: 10.1056/NEJMoa1315231. PMID 24918373
- [Derived] Mease PJ, Genovese MC, Mutebi A, Viswanathan HN, Chau D, Feng J, Erondu N, Nirula A. Improvement in Psoriasis Signs and Symptoms Assessed by the Psoriasis Symptom Inventory with Brodalumab Treatment in Patients with Psoriatic Arthritis. J Rheumatol. 2016 Feb;43(2):343-9. doi: 10.3899/jrheum.150182. Epub 2016 Jan 15. PMID 26773108
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 168 subjects were enrolled in the double-blind phase of the study. Of these 168 subjects, 156 entered the open-label extension phase (52 subjects were previously dosed with placebo, 53 subjects with brodalumab 140 mg Q2W, and 51 subjects with brodalumab 280 mg Q2W).
Groups:
- 140mg SC: 140 mg AMG 827
  AMG 827 140: 140 mg AMG 827 SC (subcutaneous)
- 280mg SC: 280 mg AMG 827
  AMG 827 280: 280 mg AMG 827 SC (subcutaneous)
- Open Label AMG 827 SC 210 or 280 mg: Open label 210 mg or 280 mg AMG 827 SC (subcutaneous), after Week 12.
Period: Placebo-controlled Phase
Arm/Group | Placebo SC | 140mg SC | 280mg SC | Open Label AMG 827 SC 210 or 280 mg
Started | 55 | 57 | 56 | 0
Completed | 52 | 53 | 51 | 0
Not Completed | 3 | 4 | 5 | 0
Period: Open-label Phase
Arm/Group | Placebo SC | 140mg SC | 280mg SC | Open Label AMG 827 SC 210 or 280 mg
Started | 0 | 0 | 0 | 156
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 156

BASELINE CHARACTERISTICS:
Population: The overall Number of Baseline Participants reflects the number of participants who continued in to the Open Label Extension Phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo SC | AMG 827 140 | AMG 827 280 | Total
Number analyzed (Participants) | 52 | 53 | 51 | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 43 | 48 | 44 | 135
  >=65 years | 9 | 5 | 7 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (13.2) | 52.8 (9.3) | 50.5 (11.8) | 52.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 33 | 36 | 97
  Male | 24 | 20 | 15 | 59

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Efficacy of AMG 827 in Psoriatic Arthritis as Measured by the Proportion of Subjects Achieving an American College of Rheumatology (ACR) 20%
Description: To evaluate the efficacy of AMG 827 in psoriatic arthritis as measured by the proportion of subjects achieving an American College of Rheumatology (ACR) 20% response at week 12. ACR20 responders are subjects with 20% improvement from baseline based off of percent changes in tender/painful joint count, swollen joint counts, physician global assessment of disease activity, and health assessment questionnaire-disability index.
Time Frame: Baseline to week 12
Population: Subjects who were randomized and had non-missing value for corresponding endpoint at the specified visit
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo SC | AMG 827 140 | AMG 827 280
Number analyzed (Participants) | 52 | 53 | 50
percentage of participants | 19.2 [9.6 to 32.5] | 39.6 [26.5 to 54] | 44 [30 to 58.7]

2. Secondary Outcome: To Evaluate the Efficacy of AMG 827 in Psoriatic Arthritis as Measured by the Proportion of Subjects Achieving an ACR 50
Description: To evaluate the efficacy of AMG 827 in psoriatic arthritis as measured by the proportion of subjects achieving an ACR 50 response at week 12. ACR50 responders are subjects with 50% improvement from baseline based off of percent changes in tender/painful joint count, swollen joint counts, physician global assessment of disease activity, and health assessment questionnaire-disability index.
Time Frame: Baseline to week 12
Population: Subjects who were randomized and had non-missing value for corresponding endpoint at the specified visit
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo SC | AMG 827 140 | AMG 827 280
Number analyzed (Participants) | 52 | 53 | 51
percentage of participants | 3.8 [0.5 to 13.2] | 15.1 [6.7 to 27.6] | 15.7 [7.0 to 28.6]

3. Secondary Outcome: To Evaluate the Efficacy of AMG 827 in Psoriatic Arthritis as Measured by the Proportion of Subjects Achieving an ACR 70
Description: To evaluate the efficacy of AMG 827 in psoriatic arthritis as measured by the proportion of subjects achieving an ACR 70 response at Week 12. ACR70 responders are subjects with 70% improvement from baseline based off of percent changes in tender/painful joint count, swollen joint counts, physician global assessment of disease activity, and health assessment questionnaire-disability index.
Time Frame: Baseline to week 12
Population: Subjects who were randomized and had non-missing value for corresponding endpoint at the specified visit
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo SC | AMG 827 140 | AMG 827 280
Number analyzed (Participants) | 52 | 53 | 51
percentage of participants | 0 [0 to 6.7] | 5.7 [1.2 to 15.7] | 5.9 [1.2 to 16.2]

4. Secondary Outcome: To Evaluate the Efficacy of AMG 827 in Psoriatic Arthritis as Measured by Change From Baseline in Clinical Disease Activity Index (CDAI)
Description: To evaluate the efficacy of AMG 827 in psoriatic arthritis as measured by Clinical Disease Activity Index (CDAI) change from baseline at week 12.
  CDAI = SJC(28) + TJC(28) + PGA + EGA
  * SJC(28): Swollen 28-Joint Count (shoulders, elbows, wrists, MCPs, PIPs including thumb IP, knees)
  * TJC(28): Tender 28-Joint Count (shoulders, elbows, wrists, MCPs, PIPs including thumb IP, knees)
  * PGA: Patient Global disease Activity (patient's self assessment of overall RA disease activity on a scale 1-10 where 10 is maximal activity) A CDAI reduction of 6.5 represents moderate improvement.
  * EGA: Evaluator's Global disease Activity (evaluator's assessment of overall RA disease activity on a scale 1-10 where 10 is maximal activity)
Time Frame: Baseline to week 12
Population: Subjects who were randomized and had non-missing value for corresponding endpoint at the specified visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo SC | AMG 827 140 | AMG 827 280
Number analyzed (Participants) | 50 | 53 | 51
score on a scale | -3.96 (10.32) | -11.32 (12.21) | -11.25 (9.16)

5. Secondary Outcome: To Evaluate the Efficacy of AMG 827 in Psoriatic Arthritis as Measured by Change From Baseline in Disease Activity Score With a 28 Joint Count (DAS 28)
Description: To evaluate the efficacy of AMG 827 in psoriatic arthritis as measured by Disease Activity Score with a 28 joint count (DAS 28) change from baseline at week 12.
  The DAS28 is a composite score derived from 4 measures. To calculate the DAS28:
  1. count the number of swollen joints (out of the 28),
  2. count the number of tender joints (out of the 28),
  3. take blood to measure the erythrocyte sedimentation rate (ESR) or C reactive protein (CRP),
  4. ask the participant to make a 'global assessment of health' (indicated by marking a 10 cm line between very good and very bad).
  These results are then fed into a complex mathematical formula to produce the overall disease activity score. A DAS28 of greater than 5.1 implies active disease, less than 3.2 low disease activity, and less than 2.6 remission.
Time Frame: Baseline to week 12
Population: Subjects who were randomized and had non-missing value for corresponding endpoint at the specified visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo SC | AMG 827 140 | AMG 827 280
Number analyzed (Participants) | 51 | 51 | 51
score on a scale | -0.42 (1.25) | -1.17 (1.39) | -1.06 (0.97)

ADVERSE EVENTS:
Groups:
- Open Label 210 mg or 280 mg AMG 827: Open label 210 mg or 280 mg AMG 827 after Week 12
Arm/Group | Placebo SC | AMG 827 140 | AMG 827 280 | Open Label 210 mg or 280 mg AMG 827
Serious Adverse Events (participants affected / at risk) | 13/52 | 15/53 | 18/51 | 31/156
Other Adverse Events (participants affected / at risk) | 52/52 | 50/53 | 50/51 | 153/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo SC (N=52) | AMG 827 140 (N=53) | AMG 827 280 (N=51) | Open Label 210 mg or 280 mg AMG 827 (N=156)
Cellulitis (Infections and infestations) | 0 | 1 | 2 | 2
Influenza (Infections and infestations) | 0 | 1 | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 1
Pnuemona (Infections and infestations) | 1 | 0 | 0 | 1
Psoas Abscess (Infections and infestations) | 1 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 1
Septic Athritis Streptococcal (Infections and infestations) | 0 | 0 | 1 | 1
Sphingomonas Paucimobilis infection (Infections and infestations) | 0 | 1 | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 3 | 0 | 2
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Coronary Artery Stenosis (Cardiac disorders) | 1 | 0 | 0 | 1
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Intervertebral Disc Protusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0 | 2
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Malignant Melinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
tendon Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Cerebral Infarction (Nervous system disorders) | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
Aortic Stenosis (Vascular disorders) | 0 | 0 | 2 | 1
Thrombosis in Device (General disorders) | 0 | 1 | 0 | 1
Diabetic Ketacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 1 | 1
Pelvi-Ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Knee Arthroplasty (Surgical and medical procedures) | 0 | 0 | 1 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo SC (N=52) | AMG 827 140 (N=53) | AMG 827 280 (N=51) | Open Label 210 mg or 280 mg AMG 827 (N=156)
Upper respiratory Tract Infection (Infections and infestations) | 8 | 14 | 11 | 33
Nasopharyngitis (Investigations) | 9 | 10 | 10 | 29
urinary tract infection (Infections and infestations) | 5 | 10 | 8 | 23
Bronchitis (Infections and infestations) | 6 | 8 | 7 | 21
Sinusitis (Infections and infestations) | 4 | 8 | 9 | 21
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 5 | 2 | 8
joint effusion (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 5
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 4
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 5
Tendon Disorder (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 3
Plantar Fascitis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 3
Spinal Osteoarthrosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 3
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2
Diarrhoea (General disorders) | 3 | 12 | 9 | 24
Nausea (Gastrointestinal disorders) | 4 | 6 | 5 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other